CLINICAL TRIAL: NCT07208799
Title: Comparison of Effectiveness of Submucosal Dexamethasone and Methylprednisolone in Management of Postoperative Sequelae in Mandibular Parasymphysis Fractures
Brief Title: Comparison of Submucosal Dexamethasone and Methylprednisolone in Postoperative Sequelae of Parasymphsis Fractures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Ammar Ali Khalid, Resident, Department of Oral and Maxillofacial Surgery / Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U1111-1329-2007
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mandible Fracture; Edema Face; Pain Management; Corticosteroid Injection
Keywords: mandible fracture; edema; pain; submucosal; dexamethasone; methylprednisolone
MeSH Terms: conditions — Mandibular Fractures; Agnosia; Edema; Pain | interventions — Dexamethasone; Methylprednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone group (Active Comparator): In this study dexamethasone sodium phosphate 8 mg (2 mL) will be administered submucosally at the surgical site 30 minutes before incision.
  Interventions: Drug: Dexamethasone
- Methylprednisolone group (Active Comparator): In this study methylprednisolone sodium succinate 40 mg (2 mL) will be administered submucosally at the surgical site 30 minutes before incision.
  Interventions: Drug: Methylprednisolone (Corticosteroid)

INTERVENTIONS:
Drug: Dexamethasone — single dose of dexamethasone 8 mg (2 mL) administered submucosally at the surgical site 30 minutes before incision.
  Arms: Dexamethasone group
Drug: Methylprednisolone (Corticosteroid) — a single dose of methylprednisolone 40 mg (2 mL) will be administered submucosally at the surgical site 30 minutes before incision.
  Arms: Methylprednisolone group

SUMMARY:
The rationale of the current research is to address the limitation of existing knowledge as it is not clear which of the two drugs (Dexamethasone or Methylprednisolone) is more effective in reduction of postoperative sequelae in patient with mandibular parasymphysis fracture. This study fills the gap by providing sound evidence on the preferred steroid option to help clinicians have more data to make decisions and improve patients' health. The result of this research will then be added to the evidence-based protocols for the treatment of parasymphysis fractures.

DETAILED DESCRIPTION:
Corticosteroids such as dexamethasone and methylprednisolone have been widely investigated in oral and maxillofacial surgery for their ability to reduce postoperative pain, edema, and trismus. Several randomized controlled trials have demonstrated significant benefit compared to placebo. For example, Hashim in 2020 reported mean VAS pain scores of 2.08 ± 0.92 with dexamethasone versus 3.43 ± 1.42 with placebo at 24 hours, and 0.50 ± 0.68 versus 2.23 ± 0.80 at 72 hours; edema scores were also lower (4.1 ± 1.43 vs. 6.0 ± 1.22 at 24 hours). Similarly, Mubeen in 2023 found that dexamethasone significantly reduced pain (2.16 ± 0.89 vs. 3.51 ± 1.23 at 24 hours) and edema (4.26 ± 1.42 vs. 5.38 ± 1.01 at 24 hours) compared to placebo in mandibular fracture patients. In contrast, Kandamani in 2022 showed that patients receiving submucosal methylprednisolone (40 mg Depomedrol) had significantly less pain, swelling, and trismus than controls at 48 and 72 hours (p < 0.05).In third molar surgery, Lim and Ngeow in 2017 observed that methylprednisolone produced significantly lower pain scores than placebo on POD 1 and 2, while dexamethasone also reduced pain but without statistical significance; both steroids, however, were equally effective in reducing swelling and trismus. Ayub and Fazal in 2022 further demonstrated that dexamethasone was superior to methylprednisolone in controlling trismus at 72 hours and swelling on postoperative days 1 and 2 (p < 0.005).

While these studies confirm the benefits of corticosteroids, none have directly compared dexamethasone and methylprednisolone in mandibular fractures, and most rely only on subjective outcomes such as VAS and facial measurements. To strengthen outcome assessment, Salgia in 2015 demonstrated that serum C-reactive protein (CRP) correlates directly with postoperative pain and inflammation, validating CRP as a reliable biomarker for quantifying the surgical inflammatory response.

To address these gaps, this double-blind randomized clinical trial will compare the effectiveness of submucosal dexamethasone (8 mg) and methylprednisolone (40 mg) in patients undergoing open reduction and internal fixation of isolated mandibular parasymphysis fractures. Pain and edema will be measured clinically at baseline, 24, and 72 hours, while serum CRP will be assessed as an objective biomarker of systemic inflammation. Analgesic consumption and adverse events will also be recorded. By combining subjective and objective outcomes, this study will provide robust evidence to guide the optimal corticosteroid choice in mandibular fracture management and contribute to evidence-based postoperative protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 40.
2. Both Gender.
3. Fracture less than a week old.
4. Isolated mandibular parasymphysis fractures.

Exclusion Criteria:

* 1. Immunocompromised patients (due to increased risk of infection and complications).

  2. Patients experiencing acute pain from conditions such as pulpitis, abscesses, or other acute infections (to ensure that acute pain does not confound the study results).

  3. Patients reporting hypersensitivity to steroids (to avoid adverse reactions).

  4. Patients taking or requiring prophylactic antibiotics or anti-inflammatory drugs before surgery (to prevent confounding effects on study outcomes).

  5. Patients with a history of systemic steroid administration for 15 days (as this could affect the study's outcomes).

  6. Patients with chronic pain problems or mental disorders (to maintain consistency in response to treatment).

  7. Patients with comminuted fractures (to maintain consistency in fracture type).

  8. Pregnant or lactating women (to avoid potential risks to the fetus and nursing infant).

  9. Smokers who smoke at least 10 cigarettes per day for 2 years (to minimize the impact of smoking on healing and recovery).

ria:

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-03 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
facial Edema | at baseline, 24 hours and 72 hours after surgery
  Edema will be assessed in millimeters via measuring tape and assessed via the 9-line method at baseline, 24 hours and 72 hours after surgery. It measures edema at 9 standardized facial landmarks bilaterally (gonion to lateral canthus, tragus to ala of the nose, tragus to commissure of the lip, tragus to midline of the chin and gonion to gonion)
pain intensity | at baseline, 24 hour and 72 hour postoperatively
  : Visual Analog Scale (VAS) will be used to evaluate the pain at the baseline, 24 hours and 72 hours after the surgery. The axis is a 10-centimeter line with the endpoints showing 0 which is no pain, and 10 which is the most severe pain. Patients will put a line where they think their pain level is, and this will be recorded

SECONDARY OUTCOMES:
serum C-reactive protein (inflammation) | baseline, 24- and 72-hours post-op
  It will be measured in mg/dL at baseline, 24- and 72-hours post-op using the hospital laboratory's standard immunoassay method.
rescue analgesia | 24 hour to 72 hour after surgery
  . Rescue analgesia will be given if VAS ≥ 4, using a fixed dose of tramadol 50 mg IV/IM (single dose). If pain persists after 6-8 hours, the same 50 mg dose may be repeated, not exceeding 400 mg in 24 hours. Total rescue analgesic consumption within 72 hours will be recorded as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dr amjad ali Bari, M.D.S (OMFS), Study Director — NISHTAR INSITUTE OF DENTISTRY, MULTAN
Locations (1):
- Nishtar Institute of Dentistry Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salgia G, Kulkarni DG, Shetty L. C-reactive protein estimation: a quantitative analysis for three nonsteroidal anti-inflammatory drugs: a randomized control trial. Indian J Dent Res. 2015 Jan-Feb;26(1):43-7. doi: 10.4103/0970-9290.156797. PMID 25961614
- [Background] Saravanan T, Balaguhan B, Venkatesh A, Geethapriya N, Goldpearlinmary, Karthick A. Prevalence of mandibular fractures. Indian J Dent Res. 2020 Nov-Dec;31(6):971-974. doi: 10.4103/ijdr.IJDR_286_18. PMID 33753671
- [Background] Singh AK, Dhungel S, Bhattarai K, Roychoudhury A. Do the Benefits of Systemic Corticosteroids Outweigh Adverse Effects During Maxillofacial Trauma Surgery? A Systematic Review and Meta-Analysis. J Oral Maxillofac Surg. 2021 Jul;79(7):1530.e1-1530.e21. doi: 10.1016/j.joms.2021.02.003. Epub 2021 Feb 9. PMID 33745861
- [Background] Nils HJ, Arce Recatala C, Castano A, Ribas D, Flores-Fraile J. Efficacy/Safety of the Use of Glucocorticoids in Oral and Maxillofacial Surgery. Dent J (Basel). 2023 Oct 17;11(10):239. doi: 10.3390/dj11100239. PMID 37886924
- [Background] Mohd YQ, Reddy S, Sinha R, Agarwal A, Fatima U, Abidullah M. Three-Dimensional Miniplate: For the Management of Mandibular Parasymphysis Fractures. Ann Maxillofac Surg. 2019 Jul-Dec;9(2):333-339. doi: 10.4103/ams.ams_172_17. PMID 31909011
- [Background] Mohamed, N.A., Hassan, R.S. & El Halawani, G. 2024. Comparison between perpendicular and conventional fixation in symphyseal and para symphyseal mandibular fractures (Randomized controlled trial). Alexandria Dental Journal.
- [Background] Kandamani J, Gouthaman SS, Ramakrishnan DS, Kumar MPS, Muthusekar MR. Evaluation of effect of submucosal administration of depomedrol in management of postoperative sequelae in mandibular fractures: A randomized clinical trial study. Natl J Maxillofac Surg. 2022 Jan-Apr;13(1):84-89. doi: 10.4103/njms.NJMS_118_20. Epub 2022 Apr 20. PMID 35911819
- [Background] Hashim, M.H., Shadab, R., Kali, B., Khan, N., Tariq, Z.R., Ali, S. and Zahid, S., 2020. Role of dexamethasone at surgical site in the control of pain and edema in the management of mandibular fracture osteosynthesis. Pakistan Oral & Dental Journal, 40(2), pp.72-75. Hunter, T.B. 2017. Fracture fixation. Radiologic Guide to Orthopedic Devices:19.
- [Background] Gadicherla S, Sasikumar P, Gill SS, Bhagania M, Kamath AT, Pentapati KC. Mandibular Fractures and Associated Factors at a Tertiary Care Hospital. Arch Trauma Res. 2016 Sep 19;5(4):e30574. doi: 10.5812/atr.30574. eCollection 2016 Dec. PMID 28144599
- [Background] Dongol A, Jaisani MR, Pradhan L, Dulal S, Sagtani A. A randomized clinical trial of the effects of submucosal dexamethasone after surgery for mandibular fractures. J Oral Maxillofac Surg. 2015 Jun;73(6):1124-32. doi: 10.1016/j.joms.2014.12.042. Epub 2015 Jan 13. PMID 25843816
- [Background] Dergin, G., Emes, Y. & Aybar, B. 2019. Evaluation and management of mandibular fracture. Trauma in dentistry. https://www.intechopen.com/chapters/65088.
- [Background] Chugh A, Singh S, Mittal Y, Chugh V. Submucosal injection of dexamethasone and methylprednisolone for the control of postoperative sequelae after third molar surgery: randomized controlled trial. Int J Oral Maxillofac Surg. 2018 Feb;47(2):228-233. doi: 10.1016/j.ijom.2017.07.009. Epub 2017 Aug 12. PMID 28811076
- [Background] Sugragan C, Sirintawat N, Kiattavornchareon S, Khoo LK, Kc K, Wongsirichat N. Do corticosteroids reduce postoperative pain following third molar intervention? J Dent Anesth Pain Med. 2020 Oct;20(5):281-291. doi: 10.17245/jdapm.2020.20.5.281. Epub 2020 Oct 30. PMID 33195806